CLINICAL TRIAL: NCT06602609
Title: Remote Acute Monitoring-based Same-day Discharge Strategy of Post Transcatheter Aortic Valve Implantation Patients Versus Standard Care at 30-Day Follow-up
Brief Title: Remote Cardiovascular Monitoring in Post-TAVI Patients
Acronym: TELE-TAVI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: King Khalid University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 24HH8773
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Aortic Valve Stenosis; Cardiac Conduction Disturbance; Digital Health; Transcatheter Aortic Valve Implantation; TAVI
Keywords: POST-TAVI; Hospital Length of Stay; Same-Day Discharge; Remote Monitoring; Ambulatory ECG; Digital Health; Valvular Heart Disease; TAVI; TAVR; Medical Device; Hospital at Home; Home Health; Telemedicine; Virtual Health; ECG; EKG; RCT; Digital Innovation; Technology; Ambulatory; Cardiology; Post-Acute; Post Acute; Digital Technology; Electrocardiogram; Clinical Trials; Telehealth; Home Telemetry
MeSH Terms: conditions — Aortic Valve Stenosis; Heart Valve Diseases

STUDY DESIGN:
Intervention Model Description: A single-centre, prospective, randomised controlled, parallel-group study with open-label randomisation concealment. A total of 216 patients will have a random assignment 1:1 into the active arm (remote monitoring) or control group (standard of care), employing computer-generated randomisation via a minimisation design based on sex and age (75 years ± 8 years).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Other): The control group adheres to the best standard of care as per current practice.
  Interventions: Other: Standard Medical Therapy
- Remote Monitoring Group (Active Comparator): Those in the remote monitoring group will be given four devices, which will help the research team make decisions about their health condition based on the data collected. The active arm group will wear the continuous ECG device for 72 hours from discharge and will be instructed to acquire a daily 12-lead ECG and record vital signs until day 7 of hospital discharge. Additionally, participants will utilise 12-lead ECG and vital signs will be measured only when experiencing symptoms.
  Interventions: Other: Remote Patient Monitoring Strategy

INTERVENTIONS:
Other: Remote Patient Monitoring Strategy — Continuous remote monitoring with the SmartCardia device includes continuous heart rate and cardiac conduction rhythm tracking through a 7-lead ECG enhanced by machine learning. This system can detect cardiac rhythm disturbances, measure breathing and heart rate, and provide live-alert notifications. Daily 12-lead ECG will be collected from each patient for 7 days after discharge; patients are instructed to perform a daily 12-lead ECG on the SHL device, along with recording blood pressure and oxygen saturation levels. Each ECG is interpreted by the trial team, and a cardiologist's interpretation is confirmed, and patients will undergo remote consultations with a cardiologist or research nurse each day if needed. During the initial 30 days of patient recruitment, if the individual exhibits potential cardiac symptoms, they can activate a remote consultation by performing an extra 12-lead ECG and recording blood pressure and oxygen saturation levels.
  Arms: Remote Monitoring Group
Other: Standard Medical Therapy — No intervention is required. Patients in this arm will fill out a self-reported anxiety report (SHAI form) and provide recent admission information
  Other Names: Current standard of care
  Arms: Control Group

SUMMARY:
The goal of this randomised clinical trial is to utilise a remote monitoring algorithm to gather essential clinical data, aiming to guide the management of post-Transcatheter Aortic Valve Implantation (TAVI) patients and reduce both postprocedural hospital length of stay and readmissions. This strategic integration of technology aims to address gaps identified in previous studies and enhance the effectiveness of post-TAVI patient care. One significant concern after TAVI is the development of heart conduction abnormalities on the ECG and abnormal rhythms, such as heart block, potentially requiring permanent pacemaker insertion. Addressing these rhythm issues is crucial for reducing the overall length of stay.

The main question it aims to answer is: Does a remote patient monitoring protocol-driven strategy reduce post-TAVI hospital length of stay and adverse events? Participants post-TAVI procedure and eligible for same-day discharge, as determined by their primary cardiologist, will be randomized upon informed consent into the active arm (remote monitoring) or control group (standard of care).

Participants in the active arm will: receive four remote monitoring devices. Receive support from a validated clinical decision-making algorithm for further management.

Participants in the control group will: adhere to the best standard of care as per current practice.

Researchers will compare the active arm to the control group to see if the remote patient monitoring protocol-driven strategy reduces post-TAVI hospital length of stay and adverse events.

DETAILED DESCRIPTION:
Given the susceptibility of post-TAVI patients to bradyarrhythmias and extended hospitalisation is not economically plausible, a shift toward remote monitoring could be both justifiable and has the potential to enhance outcomes and able to predict deterioration following TAVI. Despite the well-characterized high safety and effectiveness profile of TAVI across various surgical risk groups, the adoption of same-day discharge remains limited. Addressing post-TAVI arrhythmias is crucial to minimising the total postprocedural length of stay. Therefore, by embracing a minimalist approach and leveraging the vastly grown operators experience, the current post-TAVI care could be further enhanced with the integration of remote monitoring. This strategic shift aligns with the objective of optimising care by the ability to predict deterioration that can be treated to avoid in-hospital care.

Technology-enabled patient care and monitoring has been steadily improving, and AI-enabled remote patient monitoring devices has brought a crucial advantage to an outside-of-hospital cardiac investigation. The potential to remotely detect any adverse effects that patients might develop after the procedure is promising. There is an increased uptake of ECG telemetry, which might serve as a valuable tool that may significantly reduce hospital LOS at 30 days and possibly could reduce 3 months' adverse outcomes. This approach may enhance patient care and optimise post-TAVI outcomes through an efficient patient-tailored approach. Several studies have utilised remote or ambulatory ECG for post-TAVI on different clinical outcomes - however, to date, no RCT has been conducted using this approach. The findings of remote ECG monitoring studies are inconsistent with various monitoring periods and patient selection criteria. Although such studies utilised ECG monitoring, they did not integrate a strategy or pathway for out-of-hospital monitoring and clinical decision algorithms during home monitoring. To date, the TELE-TAVI trial will be the first monitoring study to incorporate live event detection and alert notification system supported by the bespoke Smartcardia 7-lead continuous ECG patch monitor in an RCT.

In order to better understand the impact of remote patient monitoring after TAVI, this trial proposes the utilisation of a remote monitoring algorithm to provide essential clinical data for guiding management, with the primary aim of reducing postprocedural hospital length of stay and readmissions. This strategic technology integration aims to address the gaps identified in previous studies and enhance the effectiveness of post-TAVI patient care.

Thus, it has been hypothesised that:

1. A remote patient monitoring protocol-driven strategy for same-day discharge, post-TAVI, is superior to the current standard of care follow-up in reducing cumulative 30-day hospital length of stay (LOS).
2. The novel remote patient monitoring strategy, supported by a clinical decisions algorithm, is more effective at prioritising patient presentations and optimising outcomes through early identification of adverse events, such as the need for a pacemaker, when compared to the standard of care.

The principal aims of this clinical randomised trial are:

* To facilitate a safe same-day discharge after TAVI through a remote monitoring approach in order to reduce postprocedural hospitalisation.
* To integrate an algorithm-based clinical decision-making protocol that enhances remote monitoring and the detection of post-TAVI adverse events, particularly focusing on cardiac conduction complications.
* To test the effectiveness of the remote monitoring strategy in the cost-effectiveness of post-TAVI patients' hospital admission and re-admission.

ELIGIBILITY:
Inclusion Criteria:

* Patient age must be 18 years or above.
* Post-TAVI patients without serious complications hindering same-day discharge, including vascular, neurological, and cardiac postprocedural complications necessitating inpatient care:
* Vascular: Controlled with adequate vascular hemostasis.
* Neurological: Conscious and oriented, not under the effect of residual sedation.
* Cardiac: No significant pericardial effusion.
* Elective non-emergent patient admission and nonelective cases fitting discharge criteria.
* Comfortable ambulation post-procedure.
* The patient or their caregiver must have access to a smart device.
* Ability to provide informed consent (the patient must be alert and oriented for consent).
* Adequate social support.

Exclusion Criteria:

* Hemodynamically unstable post-TAVI condition, periprocedural cardiac arrest, cerebral vascular accident, acute kidney injury (AKI) and major/life-threatening bleeding requiring blood transfusion.
* Patients with a permanent (pre-existing or new) implanted pacing device.
* Procedural failure in device delivery.
* Major vascular access complications require patients to stay.
* Inability to engage with the technology.
* Significant communication barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Estimated)
Dates: Start 2024-09-11 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Cumulative length of stay within 30 days of the procedure. | 30 days
  Post-procedural hospital length of stay will be compared between study groups

SECONDARY OUTCOMES:
The difference in rate of new PPM implantation at 3 months. | 3 months
  Difference between intervention to control groups
Rate of emergency room visits not requiring admission | 3 months
  Accident and Emergency (A&E) visits, advised by research team and unadvised
Number of all hospital admissions at 3 months | 3 months
  Planned admissions instigated by the research team vs. unplanned
Mortality Rate at 30 days | 30 days
  Mortality rate will be compared in both study groups
Patient score for the patient-reported anxiety improvement analysis | at discharge and 30 days
  Patients in both study groups will fill out the questionnaire SHAI (Short Health Anxiety Inventory) score range 3 to 38 where 38 means lower anxiety.
Number of instances of major adverse cardiovascular events | 3 months
  Major adverse cardiovascular events in this study were recognised as myocardial infarction, cerebral vascular accident (CVA), and cardiovascular-related death.

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Khamis, MBChB DIC PhD FESC FRCP, Principal Investigator — Imperial College London, Imperial College Healthcare NHS Trust
Locations (1):
- Hammersmith Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Once the study is complete and analysed, whilst individual patient results will not be disclosed, the overall research findings may be submitted for publication in a scientific journal and presented at scientific conferences following the completion of the study. A summary of the research findings will be uploaded onto the Imperial College London website. All data will be anonymised and kept confidential.

REFERENCES:
- [Background] Otto CM, Nishimura RA, Bonow RO, Carabello BA, Erwin JP 3rd, Gentile F, Jneid H, Krieger EV, Mack M, McLeod C, O'Gara PT, Rigolin VH, Sundt TM 3rd, Thompson A, Toly C. 2020 ACC/AHA Guideline for the Management of Patients With Valvular Heart Disease: A Report of the American College of Cardiology/American Heart Association Joint Committee on Clinical Practice Guidelines. Circulation. 2021 Feb 2;143(5):e72-e227. doi: 10.1161/CIR.0000000000000923. Epub 2020 Dec 17. No abstract available. PMID 33332150
- [Background] Massoullie G, Bordachar P, Irles D, Caussin C, Da Costa A, Defaye P, Jean F, Mechulan A, Mondoly P, Souteyrand G, Pereira B, Ploux S, Eschalier R. Prognosis assessment of persistent left bundle branch block after TAVI by an electrophysiological and remote monitoring risk-adapted algorithm: rationale and design of the multicentre LBBB-TAVI Study. BMJ Open. 2016 Oct 26;6(10):e010485. doi: 10.1136/bmjopen-2015-010485. PMID 27797979
- [Background] Natarajan MK, Sheth TN, Wijeysundera HC, Chavarria J, Rodes-Cabau J, Velianou JL, Radhakrishnan S, Newman T, Smith A, Wong JA, Schwalm JD, Duong M, Mian RI, Bishop MG, Healey JS. Remote ECG monitoring to reduce complications following transcatheter aortic valve implantations: the Redirect TAVI study. Europace. 2022 Oct 13;24(9):1475-1483. doi: 10.1093/europace/euac042. PMID 35699482
- [Background] Xu S, Zhang E, Qian Z, Sun J, Zou F, Wang Y, Hou X, Zou J. Mid- to Long-Term Clinical and Echocardiographic Effects of Post-procedural Permanent Pacemaker Implantation After Transcatheter Aortic Valve Replacement: A Systematic Review and Meta-Analysis. Front Cardiovasc Med. 2022 Jun 28;9:911234. doi: 10.3389/fcvm.2022.911234. eCollection 2022. PMID 35837611
- [Background] Glikson M, Nielsen JC, Kronborg MB, Michowitz Y, Auricchio A, Barbash IM, Barrabes JA, Boriani G, Braunschweig F, Brignole M, Burri H, Coats AJS, Deharo JC, Delgado V, Diller GP, Israel CW, Keren A, Knops RE, Kotecha D, Leclercq C, Merkely B, Starck C, Thylen I, Tolosana JM; ESC Scientific Document Group. 2021 ESC Guidelines on cardiac pacing and cardiac resynchronization therapy. Eur Heart J. 2021 Sep 14;42(35):3427-3520. doi: 10.1093/eurheartj/ehab364. No abstract available. PMID 34455430
- [Background] Prihadi EA, Leung M, Vollema EM, Ng ACT, Ajmone Marsan N, Bax JJ, Delgado V. Prevalence and Prognostic Relevance of Ventricular Conduction Disturbances in Patients With Aortic Stenosis. Am J Cardiol. 2017 Dec 15;120(12):2226-2232. doi: 10.1016/j.amjcard.2017.08.046. Epub 2017 Sep 18. PMID 29037444
- [Background] Muntane-Carol G, Urena M, Nombela-Franco L, Amat-Santos I, Kleiman N, Munoz-Garcia A, Atienza F, Serra V, Deyell MW, Veiga-Fernandez G, Masson JB, Canadas-Godoy V, Himbert D, Castrodeza J, Elizaga J, Francisco Pascual J, Webb JG, de la Torre Hernandez JM, Asmarats L, Pelletier-Beaumont E, Philippon F, Rodes-Cabau J. Arrhythmic burden in patients with new-onset persistent left bundle branch block after transcatheter aortic valve replacement: 2-year results of the MARE study. Europace. 2021 Feb 5;23(2):254-263. doi: 10.1093/europace/euaa213. PMID 33083813
- [Background] Hartrampf B, Jochheim D, Steffen J, Czermak T, Sadoni S, Lemmermohle E, Klier I, Estner HL, Massberg S, Mehilli J, Lackermair K, Fichtner S. Permanent pacemaker dependency in patients with new left bundle branch block and new first degree atrioventricular block after transcatheter aortic valve implantation. Sci Rep. 2021 Dec 21;11(1):24383. doi: 10.1038/s41598-021-03667-0. PMID 34934073
- [Background] Hanna G, Macdonald D, Bittira B, Horlick E, Ali N, Atoui R, Alqahtani A, Fam N, Shurrab M, Spadafore J, Allen J, Cheema A, Nalla B, Pulkkinen C, Cote S, Hennessey H, Stringer M, Leblanc S, Collin J, Fenton J, Rheault-Henry M, Lauck S, Sathananthan J, Wood D, Alnasser S. The Safety of Early Discharge Following Transcatheter Aortic Valve Implantation Among Patients in Northern Ontario and Rural Areas Utilizing the Vancouver 3M TAVI Study Clinical Pathway. CJC Open. 2022 Aug 13;4(12):1053-1059. doi: 10.1016/j.cjco.2022.08.005. eCollection 2022 Dec. PMID 36562010
- [Background] Barker M, Sathananthan J, Perdoncin E, Devireddy C, Keegan P, Grubb K, Pop AM, Depta JP, Rai D, Abtahian F, Spence MS, Mailey J, Muir DF, Russo MJ, Pineda-Salazar J, Okoh A, Smith M, Dahle TG, Rana M, Alfadhel M, Meier D, Chatfield A, Akodad M, Chuang A, Samuel R, Nestelberger T, McAlister C, Lauck S, Webb JG, Wood DA. Same-Day Discharge Post-Transcatheter Aortic Valve Replacement During the COVID-19 Pandemic: The Multicenter PROTECT TAVR Study. JACC Cardiovasc Interv. 2022 Mar 28;15(6):590-598. doi: 10.1016/j.jcin.2021.12.046. PMID 35331450
- [Background] Rosseel L, Mylotte D, Cosyns B, Vanhaverbeke M, Zweiker D, Teles RC, Angeras O, Neylon A, Rudolph TK, Wykrzykowska JJ, Patterson T, Costa G, Ojeda S, Tzikas A, Abras M, Leroux L, Van Belle E, Tchetche D, Bleiziffer S, Swaans MJ, Parma R, Blackman DJ, Van Mieghem NM, Grygier M, Redwood S, Prendergast B, Van Camp G, De Backer O. Contemporary European practice in transcatheter aortic valve implantation: results from the 2022 European TAVI Pathway Registry. Front Cardiovasc Med. 2023 Aug 14;10:1227217. doi: 10.3389/fcvm.2023.1227217. eCollection 2023. PMID 37645516
- [Background] Krishnaswamy A, Isogai T, Agrawal A, Shekhar S, Puri R, Reed GW, Yun JJ, Unai S, Burns DJP, Vargo PR, Kapadia SR. Feasibility and Safety of Same-Day Discharge Following Transfemoral Transcatheter Aortic Valve Replacement. JACC Cardiovasc Interv. 2022 Mar 28;15(6):575-589. doi: 10.1016/j.jcin.2022.01.013. PMID 35331449
- [Background] Goel A, Malik AH, Bandyopadhyay D, Chakraborty S, Gupta R, Abbott JD, Ahmad H. The 30-Day Readmission Rate of Same-Day Discharge Following Transcatheter Aortic Valve Implantation (from National Readmission Database 2015 to 2019). Am J Cardiol. 2022 Aug 1;176:112-117. doi: 10.1016/j.amjcard.2022.04.033. Epub 2022 May 27. PMID 35644697
- [Background] Panagides V, Alperi A, Mesnier J, Philippon F, Bernier M, Rodes-Cabau J. Heart failure following transcatheter aortic valve replacement. Expert Rev Cardiovasc Ther. 2021 Aug;19(8):695-709. doi: 10.1080/14779072.2021.1949987. Epub 2021 Jul 6. PMID 34227916
- [Background] Iung B, Delgado V, Rosenhek R, Price S, Prendergast B, Wendler O, De Bonis M, Tribouilloy C, Evangelista A, Bogachev-Prokophiev A, Apor A, Ince H, Laroche C, Popescu BA, Pierard L, Haude M, Hindricks G, Ruschitzka F, Windecker S, Bax JJ, Maggioni A, Vahanian A; EORP VHD II Investigators. Contemporary Presentation and Management of Valvular Heart Disease: The EURObservational Research Programme Valvular Heart Disease II Survey. Circulation. 2019 Oct;140(14):1156-1169. doi: 10.1161/CIRCULATIONAHA.119.041080. Epub 2019 Sep 12. PMID 31510787
- [Background] Nazzari H, Hawkins NM, Ezekowitz J, Lauck S, Ding L, Polderman J, Yu M, Boone RH, Cheung A, Ye J, Wood D, Webb J, Toma M. The Relationship Between Heart-Failure Hospitalization and Mortality in Patients Receiving Transcatheter Aortic Valve Replacement. Can J Cardiol. 2019 Apr;35(4):413-421. doi: 10.1016/j.cjca.2018.11.016. Epub 2018 Nov 28. PMID 30853134
- [Background] Popma JJ, Deeb GM, Yakubov SJ, Mumtaz M, Gada H, O'Hair D, Bajwa T, Heiser JC, Merhi W, Kleiman NS, Askew J, Sorajja P, Rovin J, Chetcuti SJ, Adams DH, Teirstein PS, Zorn GL 3rd, Forrest JK, Tchetche D, Resar J, Walton A, Piazza N, Ramlawi B, Robinson N, Petrossian G, Gleason TG, Oh JK, Boulware MJ, Qiao H, Mugglin AS, Reardon MJ; Evolut Low Risk Trial Investigators. Transcatheter Aortic-Valve Replacement with a Self-Expanding Valve in Low-Risk Patients. N Engl J Med. 2019 May 2;380(18):1706-1715. doi: 10.1056/NEJMoa1816885. Epub 2019 Mar 16. PMID 30883053
- [Background] Mack MJ, Leon MB, Smith CR, Miller DC, Moses JW, Tuzcu EM, Webb JG, Douglas PS, Anderson WN, Blackstone EH, Kodali SK, Makkar RR, Fontana GP, Kapadia S, Bavaria J, Hahn RT, Thourani VH, Babaliaros V, Pichard A, Herrmann HC, Brown DL, Williams M, Akin J, Davidson MJ, Svensson LG; PARTNER 1 trial investigators. 5-year outcomes of transcatheter aortic valve replacement or surgical aortic valve replacement for high surgical risk patients with aortic stenosis (PARTNER 1): a randomised controlled trial. Lancet. 2015 Jun 20;385(9986):2477-84. doi: 10.1016/S0140-6736(15)60308-7. Epub 2015 Mar 15. PMID 25788234
- [Background] VARC-3 WRITING COMMITTEE; Genereux P, Piazza N, Alu MC, Nazif T, Hahn RT, Pibarot P, Bax JJ, Leipsic JA, Blanke P, Blackstone EH, Finn MT, Kapadia S, Linke A, Mack MJ, Makkar R, Mehran R, Popma JJ, Reardon M, Rodes-Cabau J, Van Mieghem NM, Webb JG, Cohen DJ, Leon MB. Valve Academic Research Consortium 3: updated endpoint definitions for aortic valve clinical research. Eur Heart J. 2021 May 14;42(19):1825-1857. doi: 10.1093/eurheartj/ehaa799. PMID 33871579
- [Background] Vahanian A, Beyersdorf F, Praz F, Milojevic M, Baldus S, Bauersachs J, Capodanno D, Conradi L, De Bonis M, De Paulis R, Delgado V, Freemantle N, Gilard M, Haugaa KH, Jeppsson A, Juni P, Pierard L, Prendergast BD, Sadaba JR, Tribouilloy C, Wojakowski W; ESC/EACTS Scientific Document Group. 2021 ESC/EACTS Guidelines for the management of valvular heart disease. Eur Heart J. 2022 Feb 12;43(7):561-632. doi: 10.1093/eurheartj/ehab395. No abstract available. PMID 34453165
- [Background] Taylor CJ, Ordonez-Mena JM, Jones NR, Roalfe AK, Myerson SG, Prendergast BD, Hobbs FR. Survival of people with valvular heart disease in a large, English community-based cohort study. Heart. 2021 Aug;107(16):1336-1343. doi: 10.1136/heartjnl-2020-318823. Epub 2021 May 24. PMID 34031157
- [Background] Coffey S, Cairns BJ, Iung B. The modern epidemiology of heart valve disease. Heart. 2016 Jan;102(1):75-85. doi: 10.1136/heartjnl-2014-307020. Epub 2015 Nov 5. No abstract available. PMID 26541169
- [Background] Patel KP, Lim WY, Pavithran A, Assadi R, Wan D, Kennon S, Ozkor M, Earley M, Sporton S, Dhinoja M, Hayward C, Muthumala A, Hunter R, Lowe M, Lambiase P, Segal O, Mathur A, Schilling R, Baumbach A, Mullen MJ, Chow AW. Early pacemaker implantation for transcatheter aortic valve implantation is safe and effective. Pacing Clin Electrophysiol. 2022 Jan;45(1):103-110. doi: 10.1111/pace.14397. Epub 2021 Dec 26. PMID 34727374
- [Background] d'Arcy JL, Coffey S, Loudon MA, Kennedy A, Pearson-Stuttard J, Birks J, Frangou E, Farmer AJ, Mant D, Wilson J, Myerson SG, Prendergast BD. Large-scale community echocardiographic screening reveals a major burden of undiagnosed valvular heart disease in older people: the OxVALVE Population Cohort Study. Eur Heart J. 2016 Dec 14;37(47):3515-3522. doi: 10.1093/eurheartj/ehw229. Epub 2016 Jun 26. PMID 27354049